CLINICAL TRIAL: NCT03171584
Title: Comparative Study of Systemic Antifungal Drugs Used in Treatment of Onychomycosis
Brief Title: Antifungal Drugs in Treatment of Onychomycosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AMLadeed, A comparative Study of Systemic antifungal drugs used in treatment of onychomycosis, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oncho
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Antifungal Drugs in Onychomycosis
MeSH Terms: interventions — Terbinafine; Fluconazole; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Terbinafine group (Experimental): Arm (1) will receive Terbinafine (250mg/day for 6 weeks).
  Interventions: Drug: Terbinafine
- Fluconazole group (Experimental): Arm (2) will receive Fluconazole (300mg once weekly for 3monthes).
  Interventions: Drug: Terbinafine
- Itraconazole group (Experimental): Arm (3) will receive Itraconazole (400mg/day for one week per month followed by 3 free weeks ,, 2 pulses for finger nail)
  Interventions: Drug: Terbinafine

INTERVENTIONS:
Drug: Terbinafine — oral antifungal drugs
  Other Names: Fluconazole; Itraconazole

SUMMARY:
Onychomycosis refers to the fungal infection of the fingernails or toenails, caused by dermatophytes, yeast and non-dermatophyte molds that lead to distortion, discoloration, thickening and detachment from the nail bed

DETAILED DESCRIPTION:
Onychomycosis accounts for up to 30% of all superficial infections of skin and constitutes about a half of all nail abnormalities; affecting approximately 5% of population worldwide

The prevalence of onychomycosis is determined by age, social class, occupation, climate, living environment and frequency of travel Despite being common dermatological presentation, the exact prevalence of onychomycosis remains largely unknown.

Toenails are more commonly affected than fingernails due to slower rate of growth of the former, reduced blood supply and usual confinement in dark moist environments The infection is more common in adult males (particularly elderly > 60 yrs of age), diabetics, immunocompromised individuals (e.g. HIV positive), individuals with peripheral vascular (arterial) disease, previous tineapedis infection, history of trauma to the nail, or those with a family history of onychomycosis Dermatophytes whether pathogenic or saprophytes are the commonest causative nail invaders Dermatophytic onychomycosis can be divided into four major clinical types on the basis of their presenting clinical features; distal and lateral subungualonychomycosis (DLSO), proximal subungualonychomycosis (PSO), white superficial onychomycosis (WSO) and total dystrophic onychomycosis (TDO) , Among these,distal and lateral subungualonychomycosis( DLSO) is the most common form.

Clinical diagnosis by physical examination alone can be inaccurate as many non infectious conditions that mimic onychomycosis like lichen planus, psoriasis need to be ruled out . Various laboratory techniques have been used to accurately diagnose onychomycosis, with microscopy by KOH and fungal culture being the most frequently used The histopathology of nail clippings can be utilized for diagnosing onychomycosis, with periodic acid-Schiff (PAS) stain that allows easy visualization of fungal hyphae . Digital dermoscopy, also called onychoscopy, is an easy and quick procedure that allows differential diagnosis of onychomycosis from the common nail dystrophies.

Dystrophic nails can be a social impediment causing significant embarrassment that affects patient's self-esteem. In addition, thickened nails can be painful, interfere with the function of the nail unit and may cause discomfort in walking, standing and exercising.

Though initially presenting as a cosmetic problem, it can eventually lead to permanent disfigurement of the nails and serve as a source of other fungal infections . Due to these significant effects specific questionnaire was designed and validated to assess quality of life in patients with onychomycosis

Treatment is chosen depending on the modality of nail invasion, fungus species and the number of affected nails. Oral treatments are often limited by drug interactions, while topical antifungal lacquers have less efficacy . Surgery or nail debridement is another invasive treatment option in limited resistant cases .

The use of griseofulvin and ketoconazole is problematic, as there are typically high relapse rates of 50-85%. In addition, treatment must be continued for a long duration with risky systemic side effects.

Fluconazole, itraconazole and terbinafine are relatively safe antifungal drugs that have been widely used with improved treatment success, producing a mycological cure in more than 90% of fingernail infections and in about 80% of toenail infections

ELIGIBILITY:
Inclusion Criteria:

* Patients with finger nail onychomycosis of different sex and age.

Exclusion Criteria:

1. Patients taking immunosuppressive drugs or drugs affecting nail colour or growth.
2. Patients with previous trauma to the nails.
3. Pregnant and lactating women.
4. Patients with 20 nail dystrophy.
5. Patients with keratinization disorders as psoriasis and chronic medical or cutaneous diseases.
6. Patients with chronic medical or cutaneous diseases that may affect quality of life.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
cure rate of patients | one year
  Percentage of patients with complete cure in every group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Sa DC, Lamas AP, Tosti A. Oral therapy for onychomycosis: an evidence-based review. Am J Clin Dermatol. 2014 Feb;15(1):17-36. doi: 10.1007/s40257-013-0056-2. PMID 24352873
- [Result] Grover C, Khurana A. Onychomycosis: newer insights in pathogenesis and diagnosis. Indian J Dermatol Venereol Leprol. 2012 May-Jun;78(3):263-70. doi: 10.4103/0378-6323.95440. PMID 22565425
- [Result] Gupta AK, Ryder JE, Summerbell RC. Onychomycosis: classification and diagnosis. J Drugs Dermatol. 2004 Jan-Feb;3(1):51-6. PMID 14964746
- [Result] Neupane S, Pokhrel DB, Pokhrel BM. Onychomycosis: a clinico-epidemiological study. Nepal Med Coll J. 2009 Jun;11(2):92-5. PMID 19968146
- [Result] Wulkan AJ, Tosti A. Pediatric nail conditions. Clin Dermatol. 2013 Sep-Oct;31(5):564-72. doi: 10.1016/j.clindermatol.2013.06.017. PMID 24079585